CLINICAL TRIAL: NCT06328218
Title: A The Effect of Simple Gymnastics Training for Parkinson's Patients in the Community: A Preliminary Study
Brief Title: The Effect of Simple Gymnastics Training for Parkinson's Patients in the Community
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Copka Sonpashan (Other Government)
Responsible Party: Sponsor-Investigator, Copka Sonpashan, The Research Director, Chao Phya Abhaibhubejhr Hospital
Organization: Chao Phya Abhaibhubejhr Hospital (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Gymnastics ParkinsonCommunity
Record Dates: First submitted 2024-03-10; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Simple Gymnastics Training (Experimental): The elderly individuals will be arranged to undergo a continuous three-week (21 days) duration of Simple Gymnastics Training, with weekends off and training conducted only on weekdays, two sessions per day, each lasting 30 minutes. Each training session will be conducted approximately at 9.00 a.m. Apart from this,we require participants to only engage in daily activities and avoid strenuous and dangerous behaviors
  Interventions: Behavioral: Simple Gymnastics Training

INTERVENTIONS:
Behavioral: Simple Gymnastics Training — This is a simple gymnastics training that includes body swings and waist twists, as well as exercises targeting the joints in the arms and legs in various directions. It aims to help Parkinson's patients improve their physical mobility. Each training session lasts for 30 minutes, with low intensity and easy to stick to.

SUMMARY:
The goal of this clinical trial is to explore the impact of Simple Gymnastics Training on Limb motor function and mental health in Parkinson's Patients in the Community (≥60 year old) with swallowing disorders. It primarily aims to address two key aspects: 1) the prevalence of Parkinson's Diseases among community-dwelling elderly individuals, and 2) the effects of Simple Gymnastics Training on Limb motor function and mental health in community-dwelling Parkinson's Patients. All patients are required to undergo a continuous three-week (21 days) Simple Gymnastics Training, with weekends off and training conducted only on weekdays. The training will be conducted two sessions per day, lasting 30 minutes each.

DETAILED DESCRIPTION:
In the early stages of Parkinson's disease, many patients do not seek medical attention. The goal of this clinical trial is to explore the impact of Simple Gymnastics Training on Limb motor function and mental health in Parkinson's Patients in the Community (≥60 year old) with swallowing disorders. It primarily aims to address two key aspects: 1) the prevalence of Parkinson's Diseases among community-dwelling elderly individuals, and 2) the effects of Simple Gymnastics Training on Limb motor function and mental health in community-dwelling Parkinson's Patients. All patients are required to undergo a continuous three-week (21 days) Simple Gymnastics Training, with weekends off and training conducted only on weekdays. The training will be conducted two sessions per day, lasting 30 minutes each.

ELIGIBILITY:
Inclusion Criteria:

* Age >60 years.
* Meeting the diagnostic criteria for Parkinson's disease developed by the Neurology Branch of the Chinese Medical Association in 2006.

Exclusion Criteria:

* Complicated with cognitive impairment or consciousness dysfunction.
* Simultaneously suffering from severe liver, kidney failure, tumors, or hematological diseases.
* Complicated with severe liver and kidney failure, tumors, or hematological disorders.:

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Unified Parkinson's Disease Rating Scale | day 1 and day 21
  The score of the Unified Parkinson's Disease Rating Scale ranges 0 to 199 points. This assessment tool includes items such as non-motor symptoms, motor function, activities of daily living, and complications, each with corresponding scoring criteria. Higher scores reflect more severe symptoms and functional impairments. The scale is a commonly used assessment tool that can be used to evaluate the severity and progression of Parkinson's disease, as well as the effectiveness of rehabilitation treatment.

SECONDARY OUTCOMES:
The Berg Balance Scale | day 1 and day 21
  The scale consists of 14 items, each involving different balance tasks and actions such as standing, turning, walking, and more. Each item is scored based on the performance level, ranging from 0 to 4, with a maximum total score of 56. Higher scores indicate better balance ability.
Patient Health Questionnaire-9 | day 1 and day 21
  Patient Health Questionnaire-9 is a scale used to assess symptoms of depression, consisting of 9 items. Each item involves different aspects of depressive symptoms such as mood, sleep, appetite, etc. Each item is scored based on the frequency and severity of symptoms in the past two weeks, with a score range from 0 to 27. Higher scores indicate more severe symptoms. Patient Health Questionnaire-9 is widely used for screening and assessment of depression.